CLINICAL TRIAL: NCT07397819
Title: Intraperitoneal Injection of Liposomal Irinotecan as Monotherapy or in Combination With Recombinant Mutant Human Tumor Necrosis Factor or Bevacizumab for the Treatment of Malignant Ascites Following Failure of Prior Standard Therapy：A Phase Ib/II Clinical Study
Brief Title: Intraperitoneal Injection of Liposomal Irinotecan as Monotherapy or in Combination With Recombinant Mutant Human Tumor Necrosis Factor or Bevacizumab for the Treatment of Malignant Ascites Following Failure of Prior Standard Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dong sheng Zhang (Other)
Collaborators: CSPC Pharmaceutical Group Limited (Industry)
Responsible Party: Sponsor-Investigator, Dong sheng Zhang, Chief Physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2025-503-02
Record Dates: First submitted 2025-12-16; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Malignant Ascites
Keywords: Liposomal Irinotecan; Recombinant Mutant Human Tumor Necrosis Factor; Bevacizumab; Malignant Ascites; Intraperitoneal Injection
MeSH Terms: interventions — irinotecan sucrosofate; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ib Dose-Escalation Stage (Experimental)
  Interventions: Drug: liposomal irinotecan monotherapy
- Phase II Expansion Stage-ARM A (Experimental)
  Interventions: Drug: liposomal irinotecan monotherapy
- Phase II Expansion Stage-ARM B (Experimental)
  Interventions: Drug: Liposomal Irinotecan + rmhTNF-NC
- Phase II Expansion Stage-ARM C (Experimental)
  Interventions: Drug: Liposomal Irinotecan + Bevacizumab

INTERVENTIONS:
Drug: liposomal irinotecan monotherapy — A "3+3" dose-escalation design will be adopted. A total of 9-18 eligible subjects will receive liposomal irinotecan treatment, with three predefined dose levels as follows:
  Dose Level 1: 20 mg, intraperitoneal injection (ip), administered on Day 1, Day 8, Day 15, and Day 21.
  Dose Level 2: 30 mg, intraperitoneal injection (ip), administered on Day 1, Day 8, Day 15, and Day 21.
  Dose Level 3: 40 mg, intraperitoneal injection (ip), administered on Day 1, Day 8, Day 15, and Day 21.
  Each subject will receive only one treatment cycle. The dosage of liposomal irinotecan will be escalated gradually from the lowest dose level to the highest. Dose-limiting toxicities (DLT) will be monitored throughout the administration cycle. Each subject will receive only one dose level of liposomal irinotecan during the study period. All subjects will complete the relevant tests specified in the protocol during treatment to evaluate safety and preliminary efficacy. Subsequent treatment regimens will be selecte
  Arms: Phase Ib Dose-Escalation Stage
Drug: liposomal irinotecan monotherapy — Liposomal irinotecan (at RP2D, intraperitoneal injection [ip], administered on Day 1, Day 8, Day 15 and Day 21).
  Arms: Phase II Expansion Stage-ARM A
Drug: Liposomal Irinotecan + rmhTNF-NC — Liposomal Irinotecan (at RP2D dose, ip, D1, D8, D15, D21) rmhTNF-NC (300 IU per administration, ip, D1, D8, D15)
  Arms: Phase II Expansion Stage-ARM B
Drug: Liposomal Irinotecan + Bevacizumab — Liposomal Irinotecan (at RP2D dose, ip, D1, D8, D15, D21) Bevacizumab (100 mg, ip, D1, D15)
  Arms: Phase II Expansion Stage-ARM C

SUMMARY:
This study is a prospective, multi-cohort Phase Ib/II clinical trial, consisting of two stages as follows:

1. Phase Ib Dose-Escalation Stage To explore the dose-limiting toxicities (DLT) of intraperitoneally administered liposomal irinotecan in patients with malignant peritoneal effusion who have failed prior standard therapy, and to estimate the maximum tolerated dose (MTD) of the investigational agent.
2. Phase II Expansion Stage To evaluate the efficacy and safety of liposomal irinotecan as monotherapy or in combination with recombinant modified human tumor necrosis factor or bevacizumab, in the treatment of malignant peritoneal effusion in patients who have failed prior standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old, gender unrestricted.
* Histologically or cytologically confirmed malignant peritoneal effusion derived from digestive system tumors (malignancy confirmed by ascites cytology, or peritoneal metastases diagnosed clinically based on imaging findings and symptoms).
* Moderate to large volume of peritoneal effusion, with failure of initial treatment or previous intraperitoneal therapy with conventional chemotherapeutic agents and/or biological response modifiers. Moderate volume of ascites is defined as: ①Ascites depth ≥3 cm confirmed by supine abdominal ultrasound; ② Presence of clinical symptoms (chest distress, dyspnea, abdominal distension and discomfort) judged by the investigator to be related to peritoneal effusion.
* ECOG performance status score 0-2.
* Expected survival time >3 months.
* Essentially normal cardiopulmonary function.
* Adequate organ function, with subjects required to meet the following laboratory parameters:

  1. Peripheral blood count: WBC ≥4.0×10⁹/L, PLT ≥80×10⁹/L, Hb ≥90 g/L.
  2. Renal function: Serum creatinine ≤2×ULN and creatinine clearance rate (calculated by the Cockcroft-Gault formula) ≥40 ml/min.
  3. Hepatic function: Total bilirubin ≤1.5×ULN; or total bilirubin >ULN with direct bilirubin ≤ULN. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (for patients with liver metastases, ALT or AST ≤5×ULN is acceptable).
  4. Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN.
* Thyroid stimulating hormone (TSH) ≤ULN. If TSH is abnormal, serum triiodothyronine (T3) and thyroxine (T4) levels, together with clinical manifestations, shall be evaluated comprehensively; subjects in non-acute active phase are eligible for enrollment.
* For non-surgically sterilized subjects of childbearing potential or female subjects of childbearing potential: A medically approved contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) must be used during the study treatment period and for 6 months after the end of study treatment. For non-surgically sterilized female subjects of childbearing potential, serum or urine HCG test must be negative within 7 days prior to enrollment, and they must be non-lactating. For male subjects whose partners are women of childbearing potential, effective contraceptive measures must be adopted during the trial and for 6 months after the last administration of the study drug.
* Voluntarily participate in the study with good compliance, sign a written informed consent form, and be able to cooperate with follow-up assessments.

Exclusion Criteria:

* History of hypersensitivity to tumor necrosis factor (TNF), its derivative drugs, bevacizumab or its analogs, irinotecan, or liposomal irinotecan.
* Diagnosis of malignant diseases other than gastrointestinal tumors within 5 years prior to the first dose (excluding radically treated basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ).
* Receipt of any other investigational drug treatment or participation in an interventional clinical trial within 7 days prior to the first dose; or receipt of anti-tumor therapy (including Chinese herbal medicines with anti-tumor indications) within 7 days prior to the first dose of the study drug.
* Pregnant or lactating women; women of childbearing potential who are unwilling to take contraceptive measures during the study period; or men who are unwilling to use effective contraceptive measures during treatment and for 1 year thereafter.
* Significant impairment of major organ function.
* Patients with obvious bleeding tendency.
* Clinically significant or uncontrolled cardiac diseases, including unstable angina pectoris, acute myocardial infarction within 6 months prior to the first dose, New York Heart Association (NYHA) Class III/IV congestive heart failure, and uncontrolled arrhythmias (subjects with pacemakers or atrial fibrillation with well-controlled heart rate are permitted).
* Clinically significant ECG abnormalities or relevant medical history as judged by the investigator; screening QTcF interval > 480 ms. For subjects with intraventricular conduction block (QRS interval > 120 ms), JTc interval may be used instead of QTc interval (if JTc is used, it must be ≤ 340 ms).
* Uncontrolled hypertension, defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg despite optimal medical treatment; a history of hypertensive crisis or hypertensive encephalopathy.
* Severe acute infection that is uncontrolled; current fever (> 38℃), purulent or chronic infection, or unhealed wounds.
* Patients with radiologically confirmed loculated peritoneal effusion; definitely diagnosed peritoneal infection.
* Active acute or chronic hepatitis B or C infection, with hepatitis B virus (HBV) DNA > 2000 IU/mL or 10⁴ copies/mL; hepatitis C virus (HCV) RNA > 10³ copies/mL; concurrent positivity for hepatitis B surface antigen (HBsAg) and anti-HCV antibody. Subjects who have received nucleoside analog antiviral therapy and achieved viral load below the above thresholds are eligible for enrollment. A known history of human immunodeficiency virus (HIV) infection or confirmed positive HIV test results.
* Evidence or history of obvious bleeding tendency within 3 months prior to enrollment (bleeding > 30 mL within 3 months, hematemesis, melena, hematochezia); hemoptysis (> 5 mL of fresh blood within 4 weeks); a history of hereditary or acquired bleeding disorders or coagulation dysfunction. Clinically significant bleeding symptoms or definite bleeding tendency within 3 months prior to enrollment (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcer).
* A history of arterial or venous thrombotic disease within 6 weeks prior to enrollment.
* A known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Receipt of major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment, or anticipated need for major surgery during the study treatment period.
* Failure to achieve adequate recovery from toxicity and/or complications of major surgery prior to the start of treatment.
* Pregnant or lactating women; or subjects who plan to conceive or give birth during the study period from screening visit to completion of safety follow-up visit (90 days after the last dose for male subjects).
* Receipt of radiotherapy within 4 weeks prior to the first dose of study drug.
* Radiotherapy-related toxicities in subjects must have fully resolved, without the need for corticosteroid therapy, and radiation pneumonitis must be definitely excluded. For palliative radiotherapy for non-central nervous system (CNS) diseases, a 2-week washout period is permitted.
* Uncontrolled neurological or psychiatric diseases/disorders with poor compliance, resulting in inability to cooperate or report treatment responses. Uncontrolled primary brain tumors or central nervous system metastases with obvious intracranial hypertension or neuropsychiatric symptoms.
* Other conditions that, in the investigator's judgment, make the subject unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks after administration
  Defined as the highest dose at which less than 33% of subjects experience dose-limiting toxicity (DLT).
Objective Response Rate | Up to 4 weeks after the first cycle
  The proportion of subjects achieving complete response and partial response per WHO criteria.

SECONDARY OUTCOMES:
Duration of Response | from the first documentation of CR/PR to PD/death, up to 1 year
  The time interval from the first documentation of objective response in malignant ascites, to the first documentation of disease progression of ascites or death due to any cause, evaluated per the WHO criteria for malignant ascites.
Disease control rate | 4 weeks after first treatment cycle
  The proportion of subjects achieving complete response, partial response, or stable disease in malignant ascites, evaluated per the WHO criteria.
Safety and Tolerability | through study completion, an average of 1 year
  The severity of adverse events will be graded and assessed in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0,
Quality of Life | through study completion, an average of 1 year
  Assessment will be performed using the Chinese version of the Functional Assessment of Chronic Illness Therapy-Ascites Index (FACIT-AI) to evaluate the impact of malignant ascites and treatment on patients' physical function, symptom burden, and daily living ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No